CLINICAL TRIAL: NCT03757871
Title: Contribution of Acupuncture on Pain Related to the Screening of Premature Retinopathy (ROP) by Digital Camera
Acronym: ELAROP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: P171005J
Record Dates: First submitted 2018-11-13; First posted 2018-11-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-03

CONDITIONS: Laser Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser Stimulation (Experimental): laser pen acupuncture projecting an infrared beam with a wavelength of 905nm bilaterally for 30 seconds on each point.
  Interventions: Device: Laser stimulation
- Placebo (Placebo Comparator): The placebo group will have an application of the pen according to the same extinguished laser criteria.
  Interventions: Device: Laser stimulation

INTERVENTIONS:
Device: Laser stimulation — an acupuncture or placebo session will be performed 30 minutes before the fundus examination. This session will last 5 minutes.

SUMMARY:
Pain management in premature infants is essential because they are exposed to repeated minor painful procedures such as screening for premature retinopathy (ROP). Acupuncture has shown its analgesic effectiveness in many studies. Laser acupuncture is a simple, fast, side-effect-free method, but no study exists on the contribution of acupuncture in the management of pain caused by the examination of the fundus in addition to conventional therapies (suction, Glucose G30%, anaesthetic eye drops) which are not sufficiently effective.

Hypothesis: Laser acupuncture is a medical device that would reduce the pain and discomfort of premature newborns when examining the fundus with a digital camera.

DETAILED DESCRIPTION:
Randomized, single-centre, randomized, double-blind, randomized, controlled clinical trial in two parallel groups, acupuncture versus placebo as an add-on to the usual analgesic strategy (Glucose G 30%/suction and administration of a drop of anesthetic eye drops). The main objective is to evaluate the contribution of acupuncture versus placebo as an add-on to the G30% glucose solution 2 minutes before the examination associated with the instillation of a drop of oxybuprocaine administered 1 minute before the start of the examination on pain assessed at the first eye fundus (FO) by the score premature infant pain profile (PIPP) measured before the start of the examination (baseline) and on 30 seconds after the examination of both eyes.

ELIGIBILITY:
Inclusion Criteria:

* Premature from 23+0 to 30sa+6d regardless of birth weight with 1st FO for ROP screening;
* Premature birth weights < 1250g with a 1st FO for ROP screening;
* Informed consent of the holder(s) of parental authority;
* Child benefiting from a social security system

Exclusion Criteria:

* Analgesic or sedative drug treatment (benzodiazepines, morphine and related) within 48 hours of the examination.
* Known chromosomal abnormality

Ages: 23 Weeks to 31 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
score at PIPP (premature infant pain profile) ≥ 10 | 24 hours
  Measurement of pain or discomfort defined by a PIPP score ≥ 10

SECONDARY OUTCOMES:
pain and discomfort | 24 hours
  Assess pain and discomfort (score FANS). The FANS score is a validated hetero-rating scale for assessing acute newborn pain when the face is difficult to analyse. On the 0 to 10 side, the absence of pain is defined by a score < 3
heart rate variability | 24 hours
  assessment of heart rate variability (NIPE score)

CONTACTS AND LOCATIONS:
Overall Officials: Farnoux Caroline, PHD, Principal Investigator — APHP; Biran Valerie, PHD, Study Chair — APHP
Locations (1):
- Hôpital Robert Debré, Paris, France